CLINICAL TRIAL: NCT00321568
Title: An Exploratory Study on Detection of Cortical and White Matter Damage in Patients With Multiple Sclerosis Using Magnetic Resonance Imaging at 7 Tesla
Brief Title: Magnetic Resonance Imaging to Detect Brain Damage in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060154; 06-N-0154
Record Dates: First submitted 2006-05-03; First posted 2006-05-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-19

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Magnetic Resonance; MRI; Magnetic Field; MS
MeSH Terms: conditions — Multiple Sclerosis

SUMMARY:
This study will evaluate the ability of magnetic resonance imaging (MRI) using different magnet strengths (1.5, 3 and 7 Tesla) to detect damage in different parts of the brain in patients with multiple sclerosis. The higher the Tesla, the greater the ability to see brain changes. Healthy subjects will also be studied to compare findings in patients with those of normal volunteers.

Healthy normal volunteers and patients with multiple sclerosis 18-65 years of age may be eligible for this study. Patients should have minimal clinical disability. Candidates are screened with a medical history, physical examination, and blood and urine tests.

Participants undergo three MRI examinations. The first is on a 1.5 Tesla machine. The second and third - at 3 Tesla and 7 Tesla - are done within 30 days of the first. Each procedure takes about 2 hours. Before and after the 7 Tesla examination, subjects have an electrocardiogram (EKG), their blood pressure and temperature are measured and a blood sample is drawn.

MRI uses a magnetic field and radio waves to produce images of body tissues and organs. This test has several advantages over x-ray methods, such as the ability to see more clearly inside the brain and to see chemical changes that might occur in specific neurological diseases. Also, since x-rays are not used, there is no radiation risk. Radio waves are generated and changes in magnetic fields are measured and analyzed by computer. For the procedure, the subject lies on a table that is moved into a metal cylinder (the MRI scanner) that has a strong magnetic field. Earplugs are worn to muffle loud thumping noises caused by the electrical switching of the radio frequency circuits. During the MRI, subjects receive an injection of a contrast agent called Gadolinium, which brightens the images.

...

DETAILED DESCRIPTION:
OBJECTIVE: Among the factors contributing to the poor identification of grey and white matter pathology of multiple sclerosis (MS) patients, the low signal-to-noise ratio and consequential poor resolution of magnetic resonance imaging (MRI) obtained at conventional magnetic fields (i.e. 1.5 Tesla) play a significant role. Preliminary results suggest that 7T-MRI has the capability to disclose characteristics of chronic white matter lesions' heterogeneity in MS, not seen at lower field MRI. We now aim to extend those results by investigating whether lesions' heterogeneous appearance pertain not only to chronic lesions, i.e. those studied thus far, but also to newly formed lesions, i.e. those enhancing upon gadolinium injection. The latter can be identified only by imaging at 7T with contrast injection those MS patients known to already have active lesions.

STUDY POPULATION: Up to 145 patients (age range: 18-65, range in the Expanded Disability Status Scale: 0-4.5) with definite MS according to Poser criteria or other diseases of the central nervous system resembling MS from an imaging stand point and up to 120 age/gender-matched healthy volunteers will be enrolled.

DESIGN: Patients previously shown to meet both the clinical and MRI criteria for MS and an equivalent number of gender- and age-matched healthy volunteers will be studied. Initially, both patients and healthy individuals will have conventional 1.5Tesla MRI T1-weighted scans without contrast, whereas patients will also have post-contrast scans. Next, both groups of subjects will be imaged on both the 3 Tesla and 7 Tesla MRIs in a random order. In each 3 Tesla and 7 Tesla MRI study the examination will include the following sequences: 3 dimensional inversion-recovery-prepared fast spoiled gradient recalled images, 3D-fluid-attenuated inversion recovery and double inversion recovery in addition to T1 and T2 conventional weighted images.

A second group of 15 patients with or without clinical relapse who are known to be in an active stage of MS as seen by post-contrast MRI will be imaged. Each patient may undergo a standard 3T MRI within the two weeks before the 7T MRI (if needed, as no information regarding his/her disease status are otherwise available from 3T MRI performed under other NIB protocols). The former will allow ascertaining in advance his/her status of lesions activity, thus providing an adequate number of patients with active lesions imaged at 7T. Each patient may need to repeat his/her scan three times in case of magnetic instability during image acquisition. Additional 3T and 7T MRIs will be performed after 1 and 6 months to follow active lesions evolution over time.

A third group of patients with MS or any other disease of the central nervous system manifesting in magnetic resonance imaging with lesions of the white matter and grey matter which could mimic MS will be included. Each patient will undergo a 3T MRI inclusive of post-contrast sequences as well as a 7T MRI.

OUTCOME MEASURES: The number of cortical lesions as well as white matter and deep grey abnormalities will be computed on images obtained at 1.5, 3 and 7 Tesla MRIs. The study will not aim at conducting a formal comparison of cortical or white matters lesions seen on 3 Tesla and 7 Tesla. Instead, the goal is to provide preliminary information that can be used to design a formal analysis of the sensitivities of the two platforms in studying those abnormalities seen in MS. Active lesions found to be conspicuous upon contrast injection will be compared between T1 and gradient echo images at 7T. Additionally, the evolution of active lesions over time at 7T will be evaluated.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Diagnosis of MS.
  2. Age between 18 and 65.
  3. Central nervous system white matter and grey matter focal disease which may mimic MS in its imaging appearance.

EXCLUSION CRITERIA:

1. Pregnancy or breastfeeding, since contrast is harmful in people who are breastfeeding.
2. Unable to provide informed consent.
3. Permanent tattooed makeup (eyeliner, lip, etc) or general tattoos.
4. Any non-organic implant or any other device such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion device, cochlear, otologic, or ear implant, transdermal medication patch (Nitro), any metallic implants or objects, body piercing(s), bone/joint pin, screw, nail, plate, wire sutures or surgical staples, shunt.
5. Cerebral aneurysms clips, shrapnel or other metal imbedded in the body (such as from war wounds or accidents).
6. Previous work in metal fields or with machines that may have left any metallic fragments in or near the eyes.
7. Severe auto accidents in the past with non-certainty that a metal object is still present in the subject's body.
8. Any psychological contraindications for MRI (e.g., suffering from claustrophobia).

HEALTHY VOLUNTEERS INCLUSION CRITERIA:

1. Age between 18 and 65

HEALTHY VOLUNTEERS EXCLUSION CRITERIA:

1. Same as for patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-05-01; Study Completion 2011-04-19

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] BROWNELL B, HUGHES JT. The distribution of plaques in the cerebrum in multiple sclerosis. J Neurol Neurosurg Psychiatry. 1962 Nov;25(4):315-20. doi: 10.1136/jnnp.25.4.315. No abstract available. PMID 14016083
- [Background] Kidd D, Barkhof F, McConnell R, Algra PR, Allen IV, Revesz T. Cortical lesions in multiple sclerosis. Brain. 1999 Jan;122 ( Pt 1):17-26. doi: 10.1093/brain/122.1.17. PMID 10050891
- [Background] Peterson JW, Bo L, Mork S, Chang A, Trapp BD. Transected neurites, apoptotic neurons, and reduced inflammation in cortical multiple sclerosis lesions. Ann Neurol. 2001 Sep;50(3):389-400. doi: 10.1002/ana.1123. PMID 11558796